CLINICAL TRIAL: NCT06631495
Title: All-cause and Diseases-specific Mortality of High-risk HPV Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lei Li, doctor, Peking Union Medical College Hospital
Other Study IDs: HPV-ADM1
Record Dates: First submitted 2024-08-29; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-08

CONDITIONS: HPV Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HPV infection: patients with HPV infection
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — not available-observation study

SUMMARY:
The corresponding prevention strategies and treatment routes of HPV infection can be provided through investigating causes of death due to HPV infection and specialized diseases.

DETAILED DESCRIPTION:
Anxiety and panic about HPV infection have become common phenomena in tumor screening. Transitional and useless diagnosis and treatment caused by HPV infection are also common, affecting women's physical and mental health and health economic level. If the investigators can understand the causes of death related to HPV infection and specialized diseases, the investigators can provide corresponding prevention strategies and treatment routes from the level of health policies and individual methods and mechanisms, and also alleviate the related panic caused by HPV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Female participate in at least once cervical cancer screening with clear information of HPV DNA test results;
2. Having clear identification (ID number or others) that can be retrieved in the cause of death database.

Exclusion Criteria:

Cases that do not fully meet all inclusion criteria are used as exclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female participate in cervical cancer screening
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
HR-HPV infection AND all-cause and diseases-specific mortality | one year
  all-cause and diseases-specific mortality of HR-HPV infection

SECONDARY OUTCOMES:
time-period of HR-HPV infection AND all-cause and diseases-specific mortality | one year
  all-cause and diseases-specific mortality of time-period of HR-HPV infection
HR-HPV type AND all-cause and diseases-specific mortality | one year
  all-cause and diseases-specific mortality of HR-HPV type

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China